CLINICAL TRIAL: NCT00831311
Title: Phase-II Immunogenicity Study of a DTaP-IPV-Hep B-PRP~T Combined Vaccine Compared With PENTAXIM™ and ENGERIX B® PEDIATRICO at 2, 4, and 6 Months of Age in Healthy Argentinean Infants
Brief Title: Study of DTaP-IPV-Hep B-PRP~T Combined Vaccine Compared With PENTAXIM™ and ENGERIX B® PEDIATRICO in Argentinean Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3L02
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-11

CONDITIONS: Diphtheria; Tetanus; Pertussis; Haemophilus Influenzae Type b; Poliomyelitis
Keywords: Diphtheria; Tetanus; Pertussis; Whooping cough; Hepatitis B; Poliomyelitis; Haemophilus influenzae type b
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Haemophilus Infections; Poliomyelitis; Hepatitis B | interventions — DTaP-IPV-HB-PRP-T vaccine; Pentavac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DTaP IPV HB-PRP~T vaccine group
  Interventions: Biological: DTaP-IPV-HB-PRP~T
- 2 (Active Comparator): PENTAXIM™ and ENGERIX B® vaccines group
  Interventions: Biological: DTaP-IPV//PRP~T combined vaccine & Recombinant hep B vaccine

INTERVENTIONS:
Biological: DTaP-IPV-HB-PRP~T — 0.5 mL, Intramuscular
  Arms: 1
Biological: DTaP-IPV//PRP~T combined vaccine & Recombinant hep B vaccine — 0.5 mL, Intramuscular (right and left thighs, respectively)
  Other Names: PENTAXIM™; ENGERIX B® PEDIATRICO
  Arms: 2

SUMMARY:
Primary Objective:

* To demonstrate that the immune response of the DTaP-IPV-Hep B-PRP~T is non-inferior for all valences to those of the association of PENTAXIM™ and ENGERIX B® PEDIATRICO one month after a three-dose primary series.

Secondary Objectives:

* To describe in each group the immunogenicity parameters one month after the three-dose primary series.
* To describe safety profile after each vaccination in both groups.

ELIGIBILITY:
Inclusion Criteria :

* Infant of either gender, aged 50 to 70 days inclusive
* Mother is negative for HBsAg
* Born at full term of pregnancy (≥37 weeks) and with a birth weight ≥2.5 kg
* Written informed consent form signed by at least one parent or by another legal representative and an independent witness
* Parent/legal representative able to attend scheduled visits and to comply with the trial procedures during the entire duration of the trial.

Exclusion Criteria :

* Axillary temperature ≥37.1°C on the day of inclusion
* Current or planned enrolment in another clinical trial during the clinical trial period
* Known mother's history of Human Immunodeficiency Virus (HIV) infection
* Known immunodeficiency (congenital or acquired) or induced by immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy since birth, or systemic corticosteroids in the last 4 weeks (≥0.5 mg per kilogram and per day equivalent prednisolone and lasting more than 7 days)
* Receipt of blood-derived products since birth
* Acute symptoms or severe chronic illness (e.g. cardiac, renal insufficiency, diabetes, auto immune disorders, congenital defect) that may interfere with conduct or completion of trial
* Occurrence of seizures since birth
* Hypersensitivity to any of the vaccine components
* Coagulopathy contraindicating intramuscular injection
* History of (documented) clinical or serological/microbiological confirmed infection due to pertussis, tetanus, diphtheria, polio, Haemophilus influenzae type b (Hib) or hepatitis B (HB) diseases
* History of vaccination against pertussis, tetanus, diphtheria, polio, Hib or HB infections
* Vaccination within the last 4 weeks.

Ages: 50 Days to 70 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 624 (Actual)
Dates: Start 2004-10; Primary Completion 2005-11 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Córdoba, Argentina

REFERENCES:
- [Result] Tregnaghi MW, Zambrano B, Santos-Lima E. Immunogenicity and safety of an investigational hexavalent diphtheria-tetanus-acellular pertussis-inactivated poliovirus-hepatitis B-Haemophilus influenzae B conjugate combined vaccine in healthy 2-, 4-, and 6-month-old Argentinean infants. Pediatr Infect Dis J. 2011 Jun;30(6):e88-96. doi: 10.1097/INF.0b013e318212eb80. PMID 21372751
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 26 October 2004 to 10 November 2005 in 1 clinical center in Argentina.
Pre-assignment Details: A total of 624 participants who met the inclusion but no exclusion criteria were enrolled and vaccinated.
Groups:
- Group 1: DTaP-IPV-Hep B-PRP~T: Participants received 3 doses of the DTaP-IPV-Hep B-PRP~T vaccine, 1 dose each at 2, 4, and 6 months of age.
- Group 2: PENTAXIM™ and ENGERIX B®: Participants received 3 doses of PENTAXIM™ (PTaP-IPV//PRP-T) and ENGERIX B® PEDIATRICO vaccines at 2, 4, and 6 months of age.
Period: Overall Study
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B®
Started | 312 | 312
Completed | 300 | 304
Not Completed | 12 | 8
Not completed — Definitive Contraindication | 3 | 3
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B® | Total
Number analyzed (Participants) | 312 | 312 | 624
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 312 | 312 | 624
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 1.76 (0.12) | 1.77 (0.11) | 1.76 (0.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 147 | 295
  Male | 164 | 165 | 329
Region of Enrollment [Number; unit: Participants]
  Argentina | 312 | 312 | 624

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroconversion for Anti-pertussis Toxoid and Anti-filamentous Hemagglutinin Antibodies Post-vaccination With Either DTaP-IPV-Hep B-PRP~T or PENTAXIM™ and ENGERIX B®
Description: Seroconversion was assessed by means of enzyme immunoassay (EIA) for anti-pertussis toxoid (PT) and anti-filamentous hemagglutinin (FHA) antibodies. Seroconversion was defined as ≥ 4 fold increase in antibody titers from Day 0 to 30 days after the third vaccination.
Time Frame: 1 month post last vaccination
Population: Seroconversion for anti-pertussis toxoid and anti-filamentous hemagglutinin antibodies was assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Groups:
- Group 2: PENTAXIM™ and ENGERIX B®: Participants received 3 doses of PENTAXIM™ (PTaP-IPV//PRP T) and ENGERIX B® PEDIATRICO vaccines at 2, 4, and 6 months of age.
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B®
Number analyzed (Participants) | 260 | 271
Percentage of Participants
  Anti-Pertussis toxoid (N = 233, 241) | 92 | 93 [0 to 0]
  Anti-Filamentous hemagglutinin (N = 250, 249) | 93 | 90 [0 to 0]

2. Primary Outcome: Percentage of Participants With Seroprotection for Anti-Hepatitis B, Anti-Polyribosyl Ribitol Phosphate (PRP), Anti-Tetanus, Anti-Diphtheria, and Anti-Polio Antibodies After Vaccination With Either DTaP-IPV-Hep B-PRP~T or PENTAXIM™ and ENGERIX B®
Description: Immunogenicity was assessed by radioimmunoassay (RIA) for anti-hepatitis B (HBs) and anti-PRP antibodies, enzyme immunoassay (EIA) for anti-tetanus, serum neutralization (SN) for anti-diphtheria, and microneutralization for anti-polio type 1, 2, and 3 antibodies.
  Seroprotection was defined as titers ≥ 10 mIU/mL for anti-Hepatitis Bs, ≥ 0.15 μg/mL for anti-PRP, ≥ 0.01 IU/mL for anti-tetanus and anti-diphtheria, and ≥ 8 1/dil for anti-polio types 1, 2, and 3 at 30 days after the third vaccination.
Time Frame: Day 150 (1 month post-vaccination 3)
Population: Seroprotection to the vaccine antigens was assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B®
Number analyzed (Participants) | 260 | 271
Percentage of Participants
  Anti-Hepatitis B (N = 258, 271) | 99 | 100 [0 to 0]
  Anti-PRP (N = 260, 270) | 95 | 97 [0 to 0]
  Anti-Tetanus (N = 260, 271) | 100 | 100 [0 to 0]
  Anti-Diphtheria (N = 260, 271) | 100 | 100 [0 to 0]
  Anti-Polio Type 1 (N = 259, 268) | 100 | 100 [0 to 0]
  Anti-Polio Type 2 (N = 257, 269) | 100 | 100 [0 to 0]
  Anti-Polio Type 3 (N = 257, 263) | 100 | 100 [0 to 0]

3. Primary Outcome: Geometric Mean Titers of Anti-Tetanus Before and Post-vaccination With Either DTaP-IPV-Hep B-PRP~T or PENTAXIM™ and ENGERIX B®
Description: Geometric mean titers to Tetanus antigen was assessed by means of enzyme immunoassay (EIA) before the first vaccination (at Day 0) and 1 month after the third vaccination (Day 150).
Time Frame: Day 150 (1 month post-vaccination 3)
Population: Geometric mean titers to the vaccine antigens were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B®
Number analyzed (Participants) | 260 | 271
Titers
  Day 0 (N = 256, 267) | 1.14 [0.960 to 1.36] | 1.16 [0.989 to 1.37]
  Day 150 (N = 260, 271) | 2.29 [2.09 to 2.51] | 1.79 [1.66 to 1.92]

4. Primary Outcome: Geometric Mean Titers of Anti-Polio Types 1, 2, and 3 Antibodies Before and Post-vaccination With Either DTaP-IPV-Hep B-PRP~T or PENTAXIM™ and ENGERIX B®
Description: Geometric mean titers to the Polio Antigens were assessed by means of microneutralization assay for anti-polio types 1, 2, and 3 before the first vaccination (at Day 0) and 1 month post-vaccination 3 (Day 150).
Time Frame: Day 150 (1 month post-vaccination 3)
Population: Geometric mean titers to the Polio Antigens were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B®
Number analyzed (Participants) | 260 | 271
Titers
  Anti-Polio Type 1 Day 0 (N = 250, 258) | 7.41 [6.34 to 8.65] | 7.04 [6.08 to 8.15]
  Anti-Polio Type 1 Day 150 (N = 259, 268) | 4091 [3452 to 4848] | 4198 [3595 to 4901]
  Anti-Polio Type 2 Day 0 (N = 249, 261) | 11.5 [9.72 to 13.7] | 10.5 [9.02 to 12.1]
  Anti-Polio Type 2 Day 150 (N = 257, 269) | 3244 [2757 to 3817] | 3223 [2753 to 3773]
  Anti-Polio Type 3 Day 0 (N = 246, 254) | 6.89 [6.09 to 7.81] | 6.77 [6.04 to 7.60]
  Anti-Polio Type 3 Day 150 (N = 257, 263) | 3839 [3197 to 4610] | 5502 [4608 to 6570]

5. Secondary Outcome: Number of Participants Reporting At Least One Solicited Injection Site Reaction Following Each Vaccination With Either DTaP-IPV-Hep B-PRP~T or PENTAXIM™
Description: Solicited injection site reactions - erythema, edema, induration, and pain were assessed in each participant at the DTaP-IPV-Hep B-PRP~T and PENTAXIM™ injection sites
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety was assessed on the safety analysis (intent-to- treat) population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B®
Number analyzed (Participants) | 311 | 312
Participants
  Any Injection site Erythema Post-vaccination 1 | 120 | 89 [0 to 0]
  Grade 3 Erythema (≥ 5 cm) Post-vaccination 1 | 6 | 2 [0 to 0]
  Any Injection site Erythema Post-vaccination 2 | 138 | 107 [0 to 0]
  Grade 3 Erythema (≥ 5 cm) Post-vaccination 2 | 6 | 0 [0 to 0]
  Any Injection site Erythema Post-vaccination 3 | 143 | 115 [0 to 0]
  Grade 3 Erythema (≥ 5 cm) Post-vaccination 3 | 7 | 4 [0 to 0]
  Any Injection site Edema Post-vaccination 1 | 97 | 62 [0 to 0]
  Grade 3 Edema (≥ 5 cm) Post-vaccination 1 | 10 | 0 [0 to 0]
  Any Injection site Edema Post-vaccination 2 | 88 | 72 [0 to 0]
  Grade 3 Edema (≥ 5 cm) Post-vaccination 2 | 4 | 1 [0 to 0]
  Any Injection site Edema Post-vaccination 3 | 100 | 73 [0 to 0]
  Grade 3 Edema (≥ 5 cm) Post-vaccination 3 | 3 | 3 [0 to 0]
  Any Injection site Induration Post-vaccination 1 | 140 | 100 [0 to 0]
  Grade 3 Induration (≥ 5 cm) Post-vaccination 1 | 6 | 0 [0 to 0]
  Any Injection site Induration Post-vaccination 2 | 123 | 99 [0 to 0]
  Grade 3 Induration (≥ 5 cm) Post-vaccination 2 | 3 | 1 [0 to 0]
  Any Injection site Induration Post-vaccination 3 | 125 | 106 [0 to 0]
  Grade 3 Induration (≥ 5 cm) Post-vaccination 3 | 2 | 4 [0 to 0]
  Any Injection site Pain Post-vaccination 1 | 195 | 138 [0 to 0]
  Grade 3 Pain (Cries when moved) Post-vaccination 1 | 83 | 34 [0 to 0]
  Any Injection site Pain Post-vaccination 2 | 139 | 115 [0 to 0]
  Grade 3 Pain (Cries when moved) Post-vaccination 2 | 36 | 13 [0 to 0]
  Any Injection site Pain Post-vaccination 3 | 126 | 105 [0 to 0]
  Grade 3 Pain (Cries when moved) Post-vaccination 3 | 15 | 8 [0 to 0]

6. Secondary Outcome: Number of Participants Reporting At Least One Solicited Injection Site Reaction Following Each Vaccination With Either DTaP-IPV-Hep B-PRP~T or ENGERIX B®
Description: Solicited injection site reactions - erythema, edema, induration, and pain were assessed in each participant at the DTaP-IPV-Hep B-PRP~T and ENGERIX B® injection sites.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety was assessed on the safety analysis (intend-to-treat) population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B®
Number analyzed (Participants) | 311 | 312
Participants
  Any Injection site Erythema Post-vaccination 1 | 120 | 59 [0 to 0]
  Grade 3 Erythema (≥5 cm) Post-vaccination 1 | 6 | 0 [0 to 0]
  Any Injection site Erythema Post-vaccination 2 | 138 | 56 [0 to 0]
  Grade 3 Erythema (≥5 cm) Post-vaccination 2 | 6 | 1 [0 to 0]
  Any Injection site Erythema Post-vaccination 3 | 143 | 67 [0 to 0]
  Grade 3 Erythema (≥5 cm) Post-vaccination 3 | 7 | 0 [0 to 0]
  Any Injection site Edema Post-vaccination 1 | 97 | 43 [0 to 0]
  Grade 3 Edema (≥ 5 cm) Post-vaccination 1 | 10 | 0 [0 to 0]
  Any Injection site Edema Post-vaccination 2 | 88 | 37 [0 to 0]
  Grade 3 Edema (≥5 cm) Post-vaccination 2 | 4 | 0 [0 to 0]
  Any Injection site Edema Post-vaccination 3 | 100 | 42 [0 to 0]
  Grade 3 Edema (≥ 5 cm) Post-vaccination 3 | 3 | 0 [0 to 0]
  Any Injection site Induration Post-vaccination 1 | 140 | 45 [0 to 0]
  Grade 3 Induration (≥ 5 cm) Post-vaccination 1 | 6 | 0 [0 to 0]
  Any Injection site Induration Post-vaccination 2 | 123 | 41 [0 to 0]
  Grade 3 Induration (≥ 5 cm) Post-vaccination 2 | 3 | 0 [0 to 0]
  Any Injection site Induration Post-vaccination 3 | 125 | 51 [0 to 0]
  Grade 3 Induration (≥5 cm) Post-vaccination 3 | 2 | 0 [0 to 0]
  Any Injection site Pain Post-vaccination 1 | 195 | 123 [0 to 0]
  Grade 3 Pain (Cries when moved) Post-vaccination 1 | 83 | 26 [0 to 0]
  Any Injection site Pain Post-vaccination 2 | 139 | 88 [0 to 0]
  Grade 3 Pain (Cries when moved) Post-vaccination 2 | 36 | 11 [0 to 0]
  Any Injection site Pain Post-vaccination 3 | 126 | 84 [0 to 0]
  Grade 3 Pain (Cries when moved) Post-vaccination 3 | 15 | 6 [0 to 0]

7. Secondary Outcome: Number of Participants Reporting At Least One Solicited Systemic Reaction Following Vaccination With Either DTaP-IPV-Hep B-PRP~T or PENTAXIM™ and ENGERIX B®
Description: Solicited systemic reactions: Pyrexia (temperature), Somnolence, Irritability, Anorexia, Vomiting not otherwise specified (NOS), Diarrhea NOS, and Crying were assessed in each participant following vaccination.
  Grade 3 reactions defined as: Pyrexia (temperature), ≥ 39.1°C; Somnolence, sleeping most of the time; Irritability, continuously irritable for ≥ 3 hours; Anorexia, refused most or all feeds; Vomiting NOS, frequent vomiting and inability to have any oral intake; Diarrhea NOS, multiple liquid stools without any solid material; and Crying, persistent, inconsolable cry ≥ 3 hours and/or high-pitched cry.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety was assessed on the safety analysis (intent-to- treat) population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B®
Number analyzed (Participants) | 311 | 312
Participants
  Any Pyrexia Post-vaccination 1 (N = 311, 312) | 116 | 71 [0 to 0]
  Grade 3 Pyrexia Post-vaccination 1 (N = 311, 312) | 0 | 0
  Any Pyrexia Post-vaccination 2 (N = 302, 307) | 95 | 84 [0 to 0]
  Grade 3 Pyrexia Post-vaccination 2 (N = 302, 307) | 1 | 1
  Any Pyrexia Post-vaccination 3 (N = 300, 304) | 99 | 83 [0 to 0]
  Grade 3 Pyrexia Post-vaccination 3 (N = 300, 304) | 3 | 2
  Any Somnolence Post-vaccination 1 (N = 311, 312) | 143 | 109 [0 to 0]
  Grade 3 Somnolence Post-vaccination 1 (N=311, 312) | 63 | 48
  Any Somnolence Post-vaccination 2 (N = 302, 307) | 87 | 73 [0 to 0]
  Grade 3 Somnolence Post-vaccination 2 (N=302, 307) | 18 | 13
  Any Somnolence Post-vaccination 3 (N = 300, 304) | 85 | 65 [0 to 0]
  Grade 3 Somnolence Post-vaccination 3 (N=300, 304) | 22 | 14
  Any Irritability Post-vaccination 1 (N = 311, 312) | 161 | 134 [0 to 0]
  Grade 3 Irritability Post-vaccination 1; N=311,312 | 0 | 0
  Any Irritability Post-vaccination 2 (N = 302, 307) | 129 | 112 [0 to 0]
  Grade 3 Irritability Post-vaccination 2; N=302,307 | 13 | 7
  Any Irritability Post-vaccination 3 (N = 300, 304) | 115 | 97 [0 to 0]
  Grade 3 Irritability Post-vaccination 3; N=300,304 | 11 | 6
  Any Anorexia Post-vaccination 1 (N = 311, 312) | 78 | 72 [0 to 0]
  Grade 3 Anorexia Post-vaccination 1 (N = 311, 312) | 4 | 2
  Any Anorexia Post-vaccination 2 (N = 302, 307) | 68 | 52 [0 to 0]
  Grade 3 Anorexia Post-vaccination 2 (N = 302, 307) | 5 | 4
  Any Anorexia Post-vaccination 3 (N = 300, 304) | 80 | 53 [0 to 0]
  Grade 3 Anorexia Post-vaccination 3 (N = 300, 304) | 12 | 2
  Any Vomiting NOS Post-vaccination 1 (N = 311, 312) | 56 | 61 [0 to 0]
  Grade 3 Vomiting NOS Post-vaccination 1: N=311,312 | 2 | 3
  Any Vomiting NOS Post-vaccination 2 (N = 302, 307) | 34 | 41 [0 to 0]
  Grade 3 Vomiting NOS Post-vaccination 2: N=302,307 | 2 | 1
  Any Vomiting NOS Post-vaccination 3 (N = 300, 304) | 42 | 23 [0 to 0]
  Grade 3 Vomiting NOS Post-vaccination 3: N=300,304 | 2 | 0
  Any Diarrhea NOS Post-vaccination 1 (N = 311, 312) | 68 | 60 [0 to 0]
  Grade 3 Diarrhea NOS Post-vaccination 1: N=311,312 | 10 | 6
  Any Diarrhea NOS Post-vaccination 2 (N = 302, 307) | 51 | 43 [0 to 0]
  Grade 3 Diarrhea NOS Post-vaccination 2: N=302,307 | 2 | 2
  Any Diarrhea NOS Post-vaccination 3 (N = 300, 304) | 33 | 31 [0 to 0]
  Grade 3 Diarrhea NOS Post-vaccination 3: N=300,304 | 3 | 2
  Crying Post-vaccination 1 (N = 311, 312) | 152 | 113 [0 to 0]
  Grade 3 Crying Post-vaccination 1 (N = 311, 312) | 9 | 1
  Any Crying Post-vaccination 2 (N = 302, 307) | 104 | 89 [0 to 0]
  Grade 3 Crying Post-vaccination 2 (N = 302, 307) | 1 | 2
  Any Crying Post-vaccination 3 (N = 300, 304) | 78 | 71 [0 to 0]
  Grade 3 Crying Post-vaccination 3 (N = 300, 304) | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination (Day 0) up to Day 150 post-vaccination.
Arm/Group | Group 1: DTaP-IPV-Hep B-PRP~T | Group 2: PENTAXIM™ and ENGERIX B®
Serious Adverse Events (participants affected / at risk) | 19/311 | 22/312
Other Adverse Events (participants affected / at risk) | 305/311 | 307/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DTaP-IPV-Hep B-PRP~T (N=311) | Group 2: PENTAXIM™ and ENGERIX B® (N=312)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 9 (9) | 6 (6)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 3 (3)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skull Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Apnea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DTaP-IPV-Hep B-PRP~T (N=311) | Group 2: PENTAXIM™ and ENGERIX B® (N=312)
Diarrhea Not Otherwise Specified (Gastrointestinal disorders) | 119 (119) | 119 (119)
Vomiting Not Otherwise Specified (Gastrointestinal disorders) | 112 (112) | 110 (110)
Injection Site Erythemia (General disorders) | 213 (213) | 194 (194)
Injection Site Induration (General disorders) | 215 (215) | 186 (186)
Injection Site Edema (General disorders) | 172 (172) | 140 (140)
Injection Site Pain (General disorders) | 242 (242) | 202 (202)
Pyrexia (General disorders) | 209 (209) | 177 (177)
Bronchiolitis (General disorders) | 24 (24) | 27 (27)
Pharyngitis (Infections and infestations) | 23 (23) | 20 (20)
Anorexia (Metabolism and nutrition disorders) | 146 (146) | 138 (138)
Somnolence (Nervous system disorders) | 195 (195) | 156 (156)
Crying (Psychiatric disorders) | 197 (197) | 178 (178)
Irritability (Psychiatric disorders) | 218 (218) | 193 (193)
Bronchitis Not Otherwise Specified (Respiratory, thoracic and mediastinal disorders) | 33 (33) | 42 (42)
Rhinitis Not Otherwise Specified (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 28 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications